CLINICAL TRIAL: NCT06465459
Title: ESCALLE : Post-marketing Clinical Study of the LambrE System for Left Auricle Closure
Brief Title: Post-marketing Clinical Study of the LAMBRE System for Left Auricle Closure
Acronym: ESCALLE
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-A00420-47
Record Dates: First submitted 2024-05-29; First posted 2024-06-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: non-valvular atrial fibrillation; atrial fibrillation; LAMBRE system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for percutaneous left atrial closure with Lambre device implantation.
  Interventions: Procedure: LAMBRE device implantation

INTERVENTIONS:
Procedure: LAMBRE device implantation — LAMBRE device implantation

SUMMARY:
Atrial fibrillation (AF) is responsible for 15-20% of ischaemic strokes. These events are often caused by thrombus formation in the left atrium. Thromboembolic risk in AF is primarily prevented by oral anticoagulation. However, this drug-based approach has a number of limitations, the most important of which are compliance problems and, above all, the risk of haemorrhagic complications, some of which are potentially serious. Left atrial appendage closure is a therapeutic alternative for the prevention of cardioembolic risk in cases where anticoagulation is clearly contraindicated.

The CNEDiMTS opinion of 12 March 2019 defines that the LAMBRE, LIFETCH prosthesis, a device for transcatheter closure of the left atrial appendage, is authorised for the prevention of thromboembolic events in patients with non-valvular atrial fibrillation at high risk of thromboembolic events with a CHA2DS2-VASc score ≥ 4 and a formal and permanent contraindication to anticoagulants (validated by a multidisciplinary committee).

LAMBRE prosthesis in France are subject to a review of the results by the CNEDIMTS committee. Among the criteria analysed regarding the efficacy and safety of the device implantation, the result regarding the migration rate of the LAMBRE device will be one of the criteria enabling the Commission to decide on the appropriateness of the renewal of the registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a left atrial exclusion procedure according to the recommendations by the CNEDiMTS and HAS using the LAMBRE device
* Age ≥18 years
* Patient has been informed of the nature of the study and agrees to participate

Exclusion Criteria:

* Minor patient
* Patient refusing to participate in the study or unable to give informed consent (patient under guardianship, curatorship or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in cardiology departments participating in the study. Non-valvular atrial fibrillation patients at high cardio-embolic risk, contraindicated to anticoagulants, scheduled for percutaneous left atrial closure with implantation of the Lambre device will be included in the protocol and monitored as part of their care by the centers that performed the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of first cardiovascular event in patients implanted with a left atrial closure device. | during procedure and a follow-up lasting 12 months in a population having had a installation of an Lambre device
  the occurrence of one of the following events: ischaemic stroke, systemic embolism, rate of device migration and death of cardiovascular or unexplained origin occurring in patients implanted with a left atrial closure device.

SECONDARY OUTCOMES:
To evaluate the effectiveness of the device | end of procedure
  The success rate of the procedure at the end of implantation
To evaluate the effectiveness of the device | at 3 months after implantation
  the results of the scanner and/or transesophageal ultrasound concerning the rate of occlusion of the left auricle
To evaluate the effectiveness of the device | at 3 months after implantation
  the positioning of the prosthesis
To evaluate the effectiveness of the device | at 3 months after implantation
  the rate of periprosthetic shunts on the atrial side of the prosthesis
To evaluate the effectiveness of the device | at 3 months after implantation
  the rate of periprosthetic thrombus on the atrial side of the prosthesis
To evaluate the effectiveness of the device | at 1 year after implantation
  The rate of ischemic stroke
To evaluate the effectiveness of the device | at 1 year after implantation
  The rate of TIA
To evaluate the effectiveness of the device | at 1 year after implantation
  The rate of systemic embolism
To evaluate the effectiveness of the device | at 1 year after implantation
  The rate of death of cardiovascular or unexplained origin
To evaluate the effectiveness of the device | at 1 year after implantation
  The rate of death
To evaluate the effectiveness of the device | at 1 year after implantation
  The comparison of the frequency of ischemic cerebral or systemic accidents to the theoretical predicted value
To evaluate the tolerance of the procedure and the device | at the pre-discharge examination (up to 3 days)
  Complications linked or potentially linked to the implantation procedure or the device, percentage of device migration or pericardial effusion by trans-thoracic or trans-esophageal ultrasound
To evaluate the tolerance of the procedure and the device | at 3 months
  percentage of thrombosis on prosthesis or migration of the prosthesis by scanner and/or in the absence of trans-esophageal ultrasound
To evaluate the tolerance of the procedure and the device | at 1 year
  Percentage of major and/or life-threatening bleeding complications and total percentage of complications related or potentially related to the procedure or device
Description of bleeding complications not related to the device or procedure | during procedure and a follow-up lasting 12 months in a population having had a inmplantation of an Lambre device
  Percentage of patients who experienced at least one bleeding complication unrelated to the device or procedure during the entire study
Description of the population and centers | at baseline
  demographic and clinical characteristics of patients
Description of antithrombotic treatments prescribed following implantation of the device | at inclusion, at the pre-discharge examination (up to 3 days), at 30 days, 3 months and 12 months after implantation
  Percentage of patients on injectable or oral anticoagulants and on antiplatelet agents at the different follow-up times, Percentage of patients on injectable or oral anticoagulants at different follow-up times, Percentage of patients on antiplatelet agents in mono or dual therapy at the different follow-up times, Average duration of anticoagulant and antiplatelet treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier IRIART, Principal Investigator — Hôpital Cardiologique de Haut Lévêque
Locations (1):
- Hôpital Cardiologique de Haut Lévêque, Pessac, France